CLINICAL TRIAL: NCT03464097
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of Oral Ozanimod as Maintenance Therapy for Moderately to Severely Active Crohn's Disease
Brief Title: A Placebo-Controlled Study of Oral Ozanimod as Maintenance Therapy for Moderately to Severely Active Crohn's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study has terminated due to non-safety reasons; Business Objectives have changed.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPC01-3203; U1111-1203-8002 (Registry Identifier: WHO); 2023-510426-33 (Registry Identifier: EU Trial Number)
Record Dates: First submitted 2018-02-26; First posted 2018-03-13 (Actual); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease; Crohn Disease; Oral; Ozanimod; Moderately active; Severely active; RPC01; RPC01-3203
MeSH Terms: conditions — Crohn Disease | interventions — ozanimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ozanimod (Experimental)
  Interventions: Drug: Ozanimod
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ozanimod — Specified dose on specified days
  Arms: Ozanimod
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
This is a study to demonstrate the effect of oral ozanimod as maintenance therapy in participants with moderately to severely active Crohn's Disease.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit: www.BMSStudyConnect.com

Inclusion Criteria:

* Fulfilled the inclusion criteria at time of entry into the induction study and completed the week 12 efficacy assessments of the induction study
* In clinical response and/or clinical remission and/or an average daily stool frequency score ≤ 3 and an average abdominal pain score ≤ 1 with abdominal pain and stool frequency no worse than baseline at Week 12 of the Induction Study

Exclusion Criteria:

* Partial or total colectomy, small bowel resection, or an ostomy since day 1 of the induction studies or has developed a symptomatic fistula
* Had a rectal steroid therapy, rectal 5-aminosalicylates, parenteral corticosteroids, immunomodulatory agents, investigational agents or apheresis

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (765):
- United States (188):
  - Holland Center for Family Health, Peoria, Arizona
  - Local Institution - 202, Scottsdale, Arizona
  - Local Institution - 026, North Little Rock, Arkansas
  - Local Institution - 284, Camarillo, California
  - Sharp Chula Vista Medical Center, Chula Vista, California
  - Local Institution - 039, Garden Grove, California
  - Ucsd Medical Center, La Jolla, California
  - San Diego Clinical Trials, La Mesa, California
  - Local Institution - 010, Lancaster, California
  - Local Institution - 061, Los Angeles, California
  - Southern California Research Institute Medical Group, Inc., Los Angeles, California
  - Matrix Clinical Research Inc, Los Angeles, California
  - Local Institution - 110, Los Angeles, California
  - Facey Medical Foundation (Parent), Mission Hills, California
  - ABS Health, LLC, Mission Viejo, California
  - Alliance Clinical Research, Oceanside, California
  - Local Institution - 027, Orange, California
  - Palo Alto Center-Palo Alto Medical Foundation Research Institute, Palo Alto, California
  - Havana Research Institute LLC, Pasadena, California
  - Local Institution - 006, Rialto, California
  - Sutter Medical Group, Roseville, California
  - Local Institution - 280, Sacramento, California
  - Local Institution - 003, San Diego, California
  - Local Institution - 281, San Francisco, California
  - New Hope Research Development, West Covina, California
  - Local Institution - 065, Colorado Springs, Colorado
  - Local Institution - 297, Lakewood, Colorado
  - Local Institution - 182, Bristol, Connecticut
  - Local Institution - 225, Bristol, Connecticut
  - Local Institution - 091, New Haven, Connecticut
  - Local Institution - 062, Clearwater, Florida
  - Clinical Research of West Florida, Clearwater, Florida
  - South Lake Pain Institute, Clermont, Florida
  - American Research Institute Inc, Cutler Bay, Florida
  - Universal Axon Clinical Research, Doral, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - Local Institution - 218, Gainesville, Florida
  - Local Institution - 203, Hialeah, Florida
  - Floridian Clinical Research LLC, Hialeah, Florida
  - Harmony Medical Research Institute, Hialeah, Florida
  - Local Institution - 179, Hollywood, Florida
  - Vista Health Research, Homestead, Florida
  - SIH Research, Kissimmee, Florida
  - Local Institution - 016, Largo, Florida
  - Local Institution - 067, Lighthouse PT, Florida
  - Center For Advanced Gastroenterology, Maitland, Florida
  - LMG Research, Miami, Florida
  - Local Institution - 199, Miami, Florida
  - LCC Medical Research Institute, LLC, Miami, Florida
  - Local Institution - 169, Miami, Florida
  - Local Institution - 175, Miami, Florida
  - Vista Health Research, Miami, Florida
  - Local Institution - 044, Miami Springs, Florida
  - Advanced Research for Health Improvement, Naples, Florida
  - Local Institution - 192, New Port Richey, Florida
  - Local Institution - 214, New Smyrna Beach, Florida
  - Local Institution - 200, Orlando, Florida
  - Local Institution - 076, Orlando, Florida
  - Local Institution - 002, Palmetto Bay, Florida
  - Theia Clinical Research, LLC, Pinellas Park, Florida
  - Local Institution - 098, Port Orange, Florida
  - Precision Clinical Research, LLC., Sunrise, Florida
  - Local Institution - 183, Tampa, Florida
  - Apex Clinical Research, Tampa, Florida
  - Local Institution - 226, Tampa, Florida
  - Local Institution - 107, Tampa, Florida
  - Local Institution - 149, Tampa, Florida
  - Local Institution - 114, Weeki Wachee, Florida
  - Consultative Gastroenterology, Atlanta, Georgia
  - Local Institution - 037, Atlanta, Georgia
  - Local Institution - 220, Atlanta, Georgia
  - Local Institution - 222, Atlanta, Georgia
  - Local Institution - 019, Atlanta, Georgia
  - Local Institution - 063, Atlanta, Georgia
  - Local Institution - 074, Columbus, Georgia
  - Local Institution - 143, Decatur, Georgia
  - Local Institution - 028, Macon, Georgia
  - Local Institution - 115, Idaho Falls, Idaho
  - Local Institution - 194, Chicago, Illinois
  - Local Institution - 036, Chicago, Illinois
  - Local Institution - 022, Chicago, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Local Institution - 092, Evansville, Indiana
  - Local Institution - 033, Indianapolis, Indiana
  - Iowa Digestive Disease Center, Clive, Iowa
  - Local Institution - 070, Topeka, Kansas
  - Local Institution - 155, Lexington, Kentucky
  - Local Institution - 020, Baton Rouge, Louisiana
  - CroNOLA LLC, Houma, Louisiana
  - Centex Studies, Inc., Lake Charles, Louisiana
  - Clinical Trials of SW Louisiana LLC, Lake Charles, Louisiana
  - Tandem Clinical Research, LLC, Marrero, Louisiana
  - Nola Research Works, New Orleans, Louisiana
  - Local Institution - 278, Baltimore, Maryland
  - Local Institution - 129, Catonsville, Maryland
  - Local Institution - 282, Glen Burnie, Maryland
  - Local Institution - 142, Chestnut Hill, Massachusetts
  - Local Institution - 228, North Worcester, Massachusetts
  - Local Institution - 286, Springfield, Massachusetts
  - Local Institution - 024, Worcester, Massachusetts
  - Local Institution - 191, Caro, Michigan
  - Local Institution - 167, Kalamazoo, Michigan
  - Local Institution - 005, Novi, Michigan
  - Local Institution - 108, Southfield, Michigan
  - Local Institution - 301, Wyoming, Michigan
  - Local Institution - 300, Ypsilanti, Michigan
  - Local Institution - 095, Minneapolis, Minnesota
  - Local Institution - 045, Rochester, Minnesota
  - Local Institution - 274, Jackson, Mississippi
  - Local Institution - 198, Kansas City, Missouri
  - Local Institution - 029, St Louis, Missouri
  - Internal Medicine Specialists, Las Vegas, Nevada
  - Local Institution - 040, Lebanon, New Hampshire
  - Local Institution - 215, Englewood, New Jersey
  - Local Institution - 144, Brooklyn, New York
  - Local Institution - 009, Great Neck, New York
  - Local Institution - 054, Hartsdale, New York
  - Weill Cornell Medical College, New York, New York
  - Concorde Medical Group, New York, New York
  - Local Institution - 105, New York, New York
  - TrialSpark, New York, New York
  - Local Institution - 043, New York, New York
  - Local Institution - 060, North Massapequa, New York
  - Circuit Clinical, Orchard Park, New York
  - Advantage Clinical Trials, The Bronx, New York
  - Local Institution - 017, Asheville, North Carolina
  - Local Institution - 152, Charlotte, North Carolina
  - Local Institution - 055, Charlotte, North Carolina
  - Local Institution - 156, Charlotte, North Carolina
  - Local Institution - 133, Greenville, North Carolina
  - Local Institution - 302, Raleigh, North Carolina
  - Local Institution - 052, Winston-Salem, North Carolina
  - Great Lakes Medical Research, LLC, Beachwood, Ohio
  - Local Institution - 291, Cincinnati, Ohio
  - Local Institution - 018, Cleveland, Ohio
  - Local Institution - 170, Dayton, Ohio
  - Local Institution - 049, Hilliard, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - Local Institution - 141, Middleburg Heights, Ohio
  - Great Lakes Medical Research, LLC, Warren, Ohio
  - Local Institution - 087, Norman, Oklahoma
  - Local Institution - 294, Oklahoma City, Oklahoma
  - Local Institution - 208, Oklahoma City, Oklahoma
  - Local Institution - 131, Oklahoma City, Oklahoma
  - Local Institution - 185, Tulsa, Oklahoma
  - Local Institution - 217, Tulsa, Oklahoma
  - Local Institution - 113, Portland, Oregon
  - Local Institution - 197, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Penn State University Milton S Hershey Medical Center, State College, Pennsylvania
  - Local Institution - 253, Providence, Rhode Island
  - Local Institution - 289, Charleston, South Carolina
  - Local Institution - 121, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Advanced Gastroenterology, Union City, Tennessee
  - Local Institution - 158, Austin, Texas
  - Local Institution - 034, Fort Sam Houston, Texas
  - Local Institution - 056, Houston, Texas
  - Local Institution - 150, Houston, Texas
  - Biopharma Informatic Inc. Research Center, Houston, Texas
  - Centex Studies, Inc., Houston, Texas
  - GI Specialists of Houston, Houston, Texas
  - Local Institution - 303, Houston, Texas
  - Local Institution - 088, Houston, Texas
  - Local Institution - 196, Houston, Texas
  - Gulf Coast Research Group LLC, Houston, Texas
  - Accurate Clinical Research Inc, Pasadena, Texas
  - Local Institution - 071, Richardson, Texas
  - Local Institution - 085, San Antonio, Texas
  - Local Institution - 223, San Antonio, Texas
  - Local Institution - 178, San Antonio, Texas
  - Local Institution - 007, Southlake, Texas
  - Local Institution - 181, Temple, Texas
  - Local Institution - 073, Tyler, Texas
  - Local Institution - 292, Riverton, Utah
  - Local Institution - 025, Salt Lake City, Utah
  - Local Institution - 189, Gainesville, Virginia
  - Local Institution - 030, Lynchburg, Virginia
  - Local Institution - 298, Manassas, Virginia
  - Summit Clinical Research, LLC, Petersburg, Virginia
  - The Gastroenterology Group, Reston, Virginia
  - Local Institution - 072, Richmond, Virginia
  - Local Institution - 172, Roanoke, Virginia
  - Virginia Gastroenterology Institute PC, Suffolk, Virginia
  - Local Institution - 296, Williamsburg, Virginia
  - Local Institution - 125, Spokane, Washington
  - Aurora Health Care Aurora Research, Grafton, Wisconsin
  - Local Institution - 089, La Crosse, Wisconsin
- Argentina (11):
  - Local Institution - 501, Buenos Aires
  - Local Institution - 494, Buenos Aires
  - Local Institution - 571, Buenos Aires
  - Local Institution - 500, Buenos Aires
  - Local Institution - 570, Córdoba
  - Local Institution - 495, Córdoba
  - Local Institution - 569, Mar del Plata
  - Local Institution - 496, Rosario
  - Local Institution - 497, Rosario
  - Local Institution - 502, Rosario, Santa Fe
  - Local Institution - 492, San Miguel de Tucumán
- Australia (26):
  - Local Institution - 310, Concord, New South Wales
  - Local Institution - 319, Kingswood, New South Wales
  - Local Institution - 309, Liverpool, New South Wales
  - Local Institution - 318, New Lambton Heights, New South Wales
  - Local Institution - 323, Wollongong, New South Wales
  - Local Institution - 328, Herston, Queensland
  - Local Institution - 707, Maroochydore, Queensland
  - Local Institution - 313, Maroorchydore, Queensland
  - Local Institution - 321, North Mackay, Queensland
  - Local Institution - 312, South Brisbane, Queensland
  - Local Institution - 311, Woolloongabba, Queensland
  - Local Institution - 308, Adelaide, South Australia
  - Local Institution - 708, Adelaide, South Australia
  - Local Institution - 307, Bedford Park, South Australia
  - Local Institution - 326, Elizabeth Vale, South Australia
  - Local Institution - 320, Woodville South, South Australia
  - Local Institution - 317, Clayton, Victoria
  - Local Institution - 305, Fitzroy, Victoria
  - Local Institution - 329, Geelong, Victoria
  - Local Institution - 327, Melbourne, Victoria
  - Local Institution - 709, Melbourne, Victoria
  - Local Institution - 316, Murdoch, Western Australia
  - Local Institution - 315, Subiaco, Western Australia
  - Local Institution - 325, Bankstown
  - Local Institution - 330, Box Hill
  - Local Institution - 324, Sydney, NSW
- Austria (4):
  - Local Institution - 726, Innsbruck
  - Local Institution - 727, Sankt Pölten
  - Local Institution - 336, Vienna
  - Local Institution - 725, Vienna
- Belarus (2):
  - Local Institution - 745, Grodno
  - Local Institution - 737, Vitebsk
- Belgium (8):
  - Local Institution - 943, Brasschaat, Antwerpen
  - Local Institution - 940, Brussels
  - Local Institution - 939, Edegem
  - Local Institution - 937, Ghent
  - Local Institution - 942, Leuven
  - Local Institution - 936, Liège
  - Local Institution - 938, Seraing
  - Local Institution - 941, Tournai
- Bosnia and Herzegovina (4):
  - Local Institution - 743, Banja Luka
  - Local Institution - 741, Mostar
  - Local Institution - 738, Sarajevo
  - Local Institution - 742, Sarajevo
- Bulgaria (14):
  - Local Institution - 456, Blagoevgrad
  - Local Institution - 746, Plovdiv
  - Local Institution - 753, Rousse
  - Local Institution - 747, Sofia
  - Local Institution - 750, Sofia
  - Local Institution - 755, Sofia
  - Local Institution - 756, Sofia
  - Local Institution - 627, Sofia
  - Local Institution - 752, Sofia
  - Local Institution - 749, Sofia
  - Local Institution - 554, Sofia
  - Local Institution - 748, Sofia
  - Local Institution - 553, Stara Zagora
  - Local Institution - 754, Varna
- Canada (18):
  - Local Institution - 273, Calgary, Alberta
  - Local Institution - 227, Edmonton, Alberta
  - Local Institution - 269, Edmonton, Alberta
  - Local Institution - 263, Kelowna, British Columbia
  - Local Institution - 262, New Westminster, British Columbia
  - Local Institution - 255, Vancouver, British Columbia
  - Local Institution - 267, Vancouver, British Columbia
  - Local Institution - 256, Brandon, Manitoba
  - Local Institution - 261, Winnipeg, Manitoba
  - Local Institution - 268, Bridgewater, Nova Scotia
  - Local Institution - 266, Greater Sudbury, Ontario
  - Local Institution - 252, London, Ontario
  - Local Institution - 251, London, Ontario
  - Local Institution - 264, Toronto, Ontario
  - Local Institution - 257, Toronto, Ontario
  - Local Institution - 271, Vaughan, Ontario
  - Local Institution - 254, Montreal, Quebec
  - Local Institution - 270, Ottawa, Quebec
- Chile (5):
  - Local Institution - 389, Concepción
  - Local Institution - 392, Santiago
  - Local Institution - 387, Santiago
  - Local Institution - 391, Santiago
  - Local Institution - 390, Santiago
- China (36):
  - Local Institution - 423, Changzhou, Jiangsu
  - Local Institution - 369, Shanghai, Shanghai Municipality
  - Local Institution - 419, Chengdu, Sichuan
  - Local Institution - 482, Beijing
  - Local Institution - 467, Beijing
  - Local Institution - 379, Bengbu
  - Local Institution - 485, Changchun
  - Local Institution - 376, Changchun
  - Local Institution - 421, Changsha
  - Local Institution - 378, Changsha
  - Local Institution - 414, Changzhou
  - Local Institution - 422, Fuzhou
  - Local Institution - 478, Guangzhou
  - Local Institution - 472, Guangzhou
  - Local Institution - 486, Guangzhou
  - Local Institution - 470, Hangzhou, Zhejiang
  - Local Institution - 491, Hefei
  - Local Institution - 374, Kunming
  - Local Institution - 383, Luzhou
  - Local Institution - 488, Nanchang
  - Local Institution - 418, Nanjing
  - Local Institution - 375, Nanjing
  - Local Institution - 487, Nanjing
  - Local Institution - 473, Shanghai
  - Local Institution - 380, Shanghai
  - Local Institution - 377, Shanghai
  - Local Institution - 416, Shanghai
  - Local Institution - 458, Taichung City
  - Local Institution - 373, Tianjin
  - Local Institution - 475, Wuhan
  - Local Institution - 474, Wuhan
  - Local Institution - 483, Wuhan
  - Local Institution - 381, Wuxi
  - Local Institution - 415, Xi'an
  - Local Institution - 420, Xi'an
  - Local Institution - 370, Zhengzhou
- Colombia (5):
  - Local Institution - 397, Armenia, Quindío Department
  - Local Institution - 398, Barranquilla
  - Local Institution - 395, Bogotá
  - Local Institution - 396, Cali
  - Local Institution - 394, Medellín
- Croatia (6):
  - Local Institution - 453, Koprivnica
  - Local Institution - 763, Osijek
  - Local Institution - 765, Split
  - Local Institution - 452, Zagreb
  - Local Institution - 762, Zagreb
  - Local Institution - 766, Zagreb
- Czechia (12):
  - Local Institution - 767, Brno
  - Local Institution - 772, Brno
  - Local Institution - 773, Hradec Králové
  - Local Institution - 775, Most
  - Local Institution - 771, Olomouc
  - Local Institution - 774, Pardubice
  - Local Institution - 769, Pilsen
  - Local Institution - 573, Prague
  - Local Institution - 368, Prague
  - Local Institution - 776, Prague
  - Local Institution - 768, Prague
  - Local Institution - 770, Prague
- Denmark (3):
  - Local Institution - 611, Copenhagen
  - Local Institution - 610, Holbæk
  - Local Institution - 609, Nykøbing Falster
- Finland (2):
  - Local Institution - 613, Helsinki
  - Local Institution - 614, Turku
- France (18):
  - Local Institution - 647, Neuilly-sur-Seine, Cedex
  - Local Institution - 638, Amiens
  - Local Institution - 639, Béziers
  - Local Institution - 635, Blois
  - Local Institution - 634, Caen
  - Local Institution - 644, Colombes
  - Local Institution - 711, Créteil
  - Local Institution - 616, Dijon
  - Local Institution - 615, Grenoble
  - Local Institution - 633, Lillie Cedex
  - Local Institution - 646, Marseille
  - Local Institution - 507, Montpellier
  - Local Institution - 632, Nantes
  - Local Institution - 630, Pierre-Bénite
  - Local Institution - 641, Rennes
  - Local Institution - 612, Rouen
  - Local Institution - 631, Saint-Priest-en-Jarez
  - Local Institution - 643, Toulouse
- Georgia (18):
  - Local Institution - 786, Batumi
  - Local Institution - 779, Kutaisi
  - Local Institution - 248, Tbilisi
  - Local Institution - 454, Tbilisi
  - Local Institution - 783, Tbilisi
  - Local Institution - 247, Tbilisi
  - Local Institution - 778, Tbilisi
  - Local Institution - 782, Tbilisi
  - Local Institution - 552, Tbilisi
  - Local Institution - 781, Tbilisi
  - Local Institution - 793, Tbilisi
  - Local Institution - 740, Tbilisi
  - Local Institution - 784, Tbilisi
  - Local Institution - 785, Tbilisi
  - Local Institution - 335, Tbilisi
  - Local Institution - 249, Tbilisi
  - Local Institution - 455, Tbilisi
  - Local Institution - 780, Telavi
- Germany (30):
  - Local Institution - 626, Berlin
  - Local Institution - 629, Berlin
  - Local Institution - 665, Berlin
  - Local Institution - 653, Berlin
  - Local Institution - 648, Berlin
  - Local Institution - 650, Berlin
  - Local Institution - 628, Berlin
  - Local Institution - 664, Brandenburg
  - Local Institution - 732, Dachau
  - Local Institution - 662, Frankfurt
  - Local Institution - 654, Frankfurt
  - Local Institution - 574, Frankfurt am Main
  - Local Institution - 657, Frankfurt am Main
  - Local Institution - 658, Halle
  - Local Institution - 656, Halle
  - Local Institution - 659, Hamburg
  - Local Institution - 652, Hamburg
  - Local Institution - 591, Hanover
  - Local Institution - 649, Keil
  - Local Institution - 337, Leipzig
  - Local Institution - 651, Leipzig
  - Local Institution - 655, Ludwigshafen am Rhein
  - Local Institution - 730, Ludwigshafen am Rhein
  - Local Institution - 660, Mainz
  - Local Institution - 667, Münster
  - Local Institution - 620, Neuruppin
  - Local Institution - 584, Nürtingen
  - Local Institution - 661, Stuttgart
  - Local Institution - 666, Tübingen
  - Local Institution - 663, Ulm
- Greece (8):
  - Local Institution - 790, Athens
  - Local Institution - 588, Athens
  - Local Institution - 791, Athens
  - Local Institution - 792, Athens
  - Local Institution - 592, Athens, Attiki
  - Local Institution - 787, Heraklion
  - Local Institution - 789, Thessaloniki
  - Local Institution - 788, Thessaloniki
- Hong Kong (2):
  - Local Institution - 404, Hong Kong
  - Local Institution - 405, Kowloon
- Hungary (11):
  - Local Institution - 798, Békéscsaba
  - Local Institution - 803, Budapest
  - Local Institution - 804, Budapest
  - Local Institution - 556, Budapest
  - Local Institution - 801, Győr
  - Local Institution - 555, Gyula
  - Local Institution - 797, Miskolc
  - Local Institution - 800, Nagykanizsa
  - Local Institution - 816, Szekszárd
  - Local Institution - 805, Szentes
  - Local Institution - 799, Székesfehérvár
- India (11):
  - Local Institution - 444, Hyderabad, Andhra Pradesh
  - Local Institution - 407, Surat, Gujarat
  - Local Institution - 332, Gurgaon, Haryana
  - Local Institution - 445, Kochi, Kerala
  - Local Institution - 446, Ludhiana, Punjab
  - Local Institution - 443, Jaipur, Rajasthan
  - Local Institution - 399, Jaipur, Rajasthan
  - Local Institution - 408, Coimbatore, Tamil Nadu
  - Local Institution - 331, Hyderabad, Telangana
  - Local Institution - 457, Delhi
  - Local Institution - 411, New Delhi
- Ireland (2):
  - Local Institution - 975, Dublin, Dublin
  - Local Institution - 973, Dublin
- Israel (12):
  - Local Institution - 343, Afula
  - Local Institution - 345, Bat Yam
  - Local Institution - 346, Beer Jacob
  - Local Institution - 350, Haifa
  - Local Institution - 339, Jerusalem
  - Local Institution - 347, Jerusalem
  - Local Institution - 349, Kfar Saba
  - Local Institution - 344, Nahariya
  - Local Institution - 341, Petah Tikva
  - Local Institution - 342, Ramat Gan
  - Local Institution - 338, Rehovot
  - Local Institution - 340, Tel Aviv
- Italy (20):
  - Local Institution - 677, Bologna
  - Local Institution - 684, Brescia
  - Local Institution - 688, Brescia
  - Local Institution - 689, Castellana Grotte
  - Local Institution - 679, Catanzaro
  - Local Institution - 687, Chieti
  - Local Institution - 674, Messina
  - Local Institution - 672, Milan
  - Local Institution - 686, Milan
  - Local Institution - 334, Milan
  - Local Institution - 678, Monza
  - Local Institution - 685, Padua
  - Local Institution - 682, Palermo
  - Local Institution - 673, Pavia
  - Local Institution - 681, Roma
  - Local Institution - 675, Roma
  - Local Institution - 671, Rome
  - Local Institution - 680, Udine
  - Local Institution - 670, Varese
  - Local Institution - 676, Verona
- Latvia (3):
  - Local Institution - 602, Riga
  - Local Institution - 601, Riga
  - Local Institution - 600, Riga
- Lithuania (5):
  - Local Institution - 605, Kaunas
  - Local Institution - 603, Klaipėda
  - Local Institution - 607, Vilnius
  - Local Institution - 606, Vilnius
  - Local Institution - 604, Vilnius
- Mexico (10):
  - Local Institution - 526, Zapapan, Jalisco
  - Local Institution - 532, Monterrey, Nuevo León
  - Local Institution - 525, Monterrey, Nuevo León
  - Local Institution - 447, Monterrey, Nuevo León
  - Local Institution - 449, Monterrey, Nuevo León
  - Local Institution - 529, Querétaro City, Querétaro
  - Local Institution - 528, Chihuahua City
  - Local Institution - 448, Mexico City
  - Local Institution - 527, México
  - Local Institution - 530, Tlalpan
- Moldova (4):
  - Local Institution - 811, Chisinau
  - Local Institution - 809, Chisinau
  - Local Institution - 812, Chisinau
  - Local Institution - 813, Chisinau
- Netherlands (6):
  - Local Institution - 952, Amsterdam
  - Local Institution - 955, Amsterdam
  - Local Institution - 956, Groningen
  - Local Institution - 949, Nijmegen
  - Local Institution - 951, Sittard-Geleen
  - Local Institution - 954, Tilburg
- Poland (55):
  - Local Institution - 403, Zamość, Lublin Voivodeship
  - Local Institution - 597, Zamość, Lublin Voivodeship
  - Local Institution - 820, Bialystok
  - Local Institution - 818, Bochnia
  - Local Institution - 580, Częstochowa
  - Local Institution - 988, Elblag
  - Local Institution - 579, Gdansk
  - Local Institution - 978, Gdansk
  - Local Institution - 577, Gdynia
  - Local Institution - 906, Jelenia Góra
  - Local Institution - 757, Józefów
  - Local Institution - 238, Katowice
  - Local Institution - 578, Katowice
  - Local Institution - 828, Katowice
  - Local Institution - 819, Katowice
  - Local Institution - 815, Krakow
  - Local Institution - 823, Krakow
  - Local Institution - 826, Krakow
  - Local Institution - 834, Ksawerów
  - Local Institution - 817, Kłodzko
  - Local Institution - 581, Lodz
  - Local Institution - 829, Lodz
  - Local Institution - 888, Lodz
  - Local Institution - 981, Lodz
  - Local Institution - 760, Lublin
  - Local Institution - 976, Nowy Targ
  - Local Institution - 830, Olsztyn
  - Local Institution - 402, Opole
  - Local Institution - 400, Oświęcim
  - Local Institution - 758, Poznan
  - Local Institution - 575, Poznan
  - Local Institution - 401, Poznan
  - Local Institution - 963, Rzeszów
  - Local Institution - 979, Sopot
  - Local Institution - 239, Sopot
  - Local Institution - 835, Szczecin
  - Local Institution - 235, Szczecin
  - Local Institution - 822, Torun
  - Local Institution - 824, Tychy
  - Local Institution - 827, Ul. Piotrkowska 177
  - Local Institution - 410, Warsaw
  - Local Institution - 576, Warsaw
  - Local Institution - 833, Warsaw
  - Local Institution - 989, Warsaw
  - Local Institution - 236, Warsaw
  - Local Institution - 586, Warsaw
  - Local Institution - 807, Warsaw
  - Local Institution - 893, Wierzchosławice
  - Local Institution - 983, Wroclaw
  - Local Institution - 984, Wroclaw
  - Local Institution - 582, Wroclaw
  - Local Institution - 982, Wroclaw
  - Local Institution - 831, Wroclaw
  - Local Institution - 987, Wroclaw
  - Local Institution - 832, Wroclaw
- Portugal (4):
  - Local Institution - 959, Coimbra
  - Local Institution - 958, Guimarães
  - Local Institution - 961, Loures
  - Local Institution - 957, Viana do Castelo
- Romania (10):
  - Local Institution - 808, Bucharest
  - Local Institution - 836, Bucharest
  - Local Institution - 499, Bucharest
  - Local Institution - 795, Bucharest
  - Local Institution - 837, Bucharest
  - Local Institution - 839, Bucharest
  - Local Institution - 842, Bucharest
  - Local Institution - 838, Cluj-Napoca
  - Local Institution - 843, Craiova
  - Local Institution - 840, Târgu Mureş
- Russia (53):
  - Local Institution - 871, Barnaul
  - Local Institution - 589, Bataysk
  - Local Institution - 621, Chelyabinsk
  - Local Institution - 991, Chelyabinsk
  - Local Institution - 598, Chita
  - Local Institution - 848, Irkutsk
  - Local Institution - 998, Kaliningrad
  - Local Institution - 882, Kaluga
  - Local Institution - 892, Kazan'
  - Local Institution - 849, Kemerovo
  - Local Institution - 599, Khanty-Mansiysk
  - Local Institution - 927, Krasnoyarsk
  - Local Institution - 566, Moscow
  - Local Institution - 851, Moscow
  - Local Institution - 873, Moscow
  - Local Institution - 870, Moscow
  - Local Institution - 869, Moscow
  - Local Institution - 990, Nizhny Novgorod
  - Local Institution - 594, Novosibirsk
  - Local Institution - 853, Novosibirsk
  - Local Institution - 876, Novosibirsk
  - Local Institution - 996, Omsk
  - Local Institution - 875, Orenburg
  - Local Institution - 867, Penza
  - Local Institution - 858, Petrozavodsk
  - Local Institution - 859, Pushkin
  - Local Institution - 960, Pyatigorsk
  - Local Institution - 846, Pyatigorsk
  - Local Institution - 863, Saint Petersburg
  - Local Institution - 993, Saint Petersburg
  - Local Institution - 862, Saint Petersburg
  - Local Institution - 868, Saint Petersburg
  - Local Institution - 847, Saint Petersburg
  - Local Institution - 857, Saint Petersburg
  - Local Institution - 845, Saint Petersburg
  - Local Institution - 856, Saint Petersburg
  - Local Institution - 879, Saint Petersburg
  - Local Institution - 878, Saint Petersburg
  - Local Institution - 874, Saint Petersburg
  - Local Institution - 865, Samara
  - Local Institution - 844, Samara
  - Local Institution - 866, Sochi
  - Local Institution - 877, Tomsk
  - Local Institution - 806, Tula
  - Local Institution - 881, Ufa
  - Local Institution - 861, Ufa
  - Local Institution - 855, Veliky Novgorod
  - Local Institution - 935, Vladimir
  - Local Institution - 999, Vladivostok
  - Local Institution - 986, Vladivostok
  - Local Institution - 880, Volgograd
  - Local Institution - 583, Yekaterinburg
  - Local Institution - 872, Yekaterinburg
- Saudi Arabia (4):
  - Local Institution - 534, Dammam
  - Local Institution - 537, Jeddah
  - Local Institution - 536, Riyadh
  - Local Institution - 535, Riyadh
- Local Institution - 546, Cape Town, Senegal
- Serbia (12):
  - Local Institution - 241, Belgrade
  - Local Institution - 245, Belgrade
  - Local Institution - 887, Belgrade
  - Local Institution - 246, Belgrade
  - Local Institution - 596, Belgrade
  - Local Institution - 886, Belgrade
  - Local Institution - 890, Belgrade
  - Local Institution - 891, Kragujevac
  - Local Institution - 884, Novi Sad
  - Local Institution - 885, Pančevo
  - Local Institution - 585, Vršac
  - Local Institution - 889, Zrenjanin
- Slovakia (7):
  - Local Institution - 900, Bratislava
  - Local Institution - 894, Bratislava
  - Local Institution - 895, Brezno
  - Local Institution - 899, Nitra
  - Local Institution - 897, Nové Zámky
  - Local Institution - 898, Prešov
  - Local Institution - 896, Rimavská Sobota
- Local Institution - 904, Celje, Slovenia
- South Africa (7):
  - Local Institution - 543, Gauteng
  - Local Institution - 545, Kempton Park
  - Local Institution - 544, Pretoria
  - Local Institution - 542, Pretoria
  - Local Institution - 549, Pretoria
  - Local Institution - 548, Somerset West
  - Local Institution - 547, Val de Grace
- South Korea (15):
  - Local Institution - 437, Ansan
  - Local Institution - 441, Busan
  - Local Institution - 434, Busan
  - Local Institution - 431, Busan
  - Local Institution - 432, Daegu
  - Local Institution - 435, Guri-si
  - Local Institution - 436, Seongnam-si
  - Local Institution - 433, Seoul
  - Local Institution - 440, Seoul
  - Local Institution - 430, Seoul
  - Local Institution - 442, Seoul
  - Local Institution - 438, Seoul
  - Local Institution - 427, Seoul
  - Local Institution - 439, Seoul
  - Local Institution - 429, Suwon
- Spain (16):
  - Local Institution - 703, Alicante
  - Local Institution - 690, Badalona
  - Local Institution - 694, Barcelona
  - Local Institution - 702, Córdoba
  - Local Institution - 699, Girona
  - Local Institution - 701, Las Palmas de Gran Canaria
  - Local Institution - 691, Madrid
  - Local Institution - 695, Madrid
  - Local Institution - 692, Madrid
  - Local Institution - 693, Majadahonda, Madrid
  - Local Institution - 698, San Cristóbal de La Laguna
  - Local Institution - 706, Santander
  - Local Institution - 696, Seville
  - Local Institution - 705, Seville
  - Local Institution - 697, Valencia
  - Local Institution - 700, Viladecans
- Local Institution - 625, Stockholm, Sweden
- Switzerland (3):
  - Local Institution - 967, Bern
  - Local Institution - 968, Sankt Gallen
  - Local Institution - 969, Zurich
- Taiwan (8):
  - Local Institution - 460, Kaohsiung City
  - Local Institution - 463, Kaohsiung, San Ming Dist.
  - Local Institution - 363, Kozlu
  - Local Institution - 461, Niao-Sung Hsiang Kaohsiung County
  - Local Institution - 459, Tainan, Taiana
  - Local Institution - 462, Taoyuan
  - Local Institution - 464, Tapei, Beitou Dist.
  - Local Institution - 465, Tapei
- Turkey (Türkiye) (11):
  - Local Institution - 357, Ankara
  - Local Institution - 356, Ankara
  - Local Institution - 360, Bursa
  - Local Institution - 365, Elâzığ
  - Local Institution - 362, Istanbul
  - Local Institution - 358, Istanbul
  - Local Institution - 361, Istanbul
  - Local Institution - 355, Istanbul
  - Local Institution - 354, Izmit/Kocaeli
  - Local Institution - 353, Kadiköy/Istanbul
  - Local Institution - 359, Trabzon
- Ukraine (38):
  - Local Institution - 914, Chernivtsi
  - Local Institution - 922, Chernivtsi
  - Local Institution - 950, Dnipropetrovsk
  - Local Institution - 229, Ivano-Frankivsk
  - Local Institution - 929, Ivano-Frankivsk
  - Local Institution - 912, Ivano-Frankivsk
  - Local Institution - 919, Kharkiv
  - Local Institution - 965, Kharkiv
  - Local Institution - 920, Khmelnytskyi
  - Local Institution - 933, Kropyvnytskyi
  - Local Institution - 901, Kyiv
  - Local Institution - 923, Kyiv
  - Local Institution - 915, Kyiv
  - Local Institution - 243, Kyiv
  - Local Institution - 563, Kyiv
  - Local Institution - 911, Kyiv
  - Local Institution - 244, Kyiv
  - Local Institution - 564, Kyiv
  - Local Institution - 918, Kyiv
  - Local Institution - 908, Kyiv
  - Local Institution - 977, Kyiv
  - Local Institution - 562, Kyiv
  - Local Institution - 240, Lutsk
  - Local Institution - 590, Lutsk
  - Local Institution - 234, Lviv
  - Local Institution - 974, Lviv
  - Local Institution - 910, Lviv
  - Local Institution - 242, Odesa
  - Local Institution - 902, Odesa
  - Local Institution - 905, Poltava
  - Local Institution - 934, Ternopil
  - Local Institution - 909, Vinnytsia
  - Local Institution - 932, Vinnytsia
  - Local Institution - 224, Vinnytsia
  - Local Institution - 924, Vinnytsia
  - Local Institution - 971, Vinnytsia
  - Local Institution - 587, Zaporizhia
  - Local Institution - 925, Zaporizhzhya
- United Kingdom (15):
  - Local Institution - 723, Southampton, Hampshire
  - Local Institution - 729, London, LND
  - Local Institution - 557, Birmingham
  - Local Institution - 714, Bristol
  - Local Institution - 560, Cardiff
  - Local Institution - 558, Chorley
  - Local Institution - 559, Corbridge Road
  - Local Institution - 712, Dundonald
  - Local Institution - 713, Glasgow
  - Local Institution - 716, Lancashire Blackpool
  - Local Institution - 722, London
  - Local Institution - 715, London
  - Local Institution - 561, North Manchester Science Park
  - Local Institution - 593, Shrewsbury
  - Local Institution - 718, Torquay

REFERENCES:
- [Derived] Feagan BG, Schreiber S, Afzali A, Rieder F, Hyams J, Kollengode K, Pearlman J, Son V, Marta C, Wolf DC, D'Haens GG. Ozanimod as a novel oral small molecule therapy for the treatment of Crohn's disease: The YELLOWSTONE clinical trial program. Contemp Clin Trials. 2022 Nov;122:106958. doi: 10.1016/j.cct.2022.106958. Epub 2022 Oct 5. PMID 36208720
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/home

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a maintenance study.
Pre-assignment Details: Participants who completed initial 12 weeks of treatment in induction studies RPC01-3201 (NCT03440372) or RPC01-3202 (NCT03440385) and are in clinical response (CDAI [Crohn's Disease Activity Index] reduction from baseline ≥100 points or CDAI score<150),clinical remission (CDAI score < 150),and/or have an average daily stool frequency score ≤ 3 and an average abdominal pain score ≤1with abdominal pain and stool frequency no worse than baseline were eligible to participate.
Groups:
- Ozanimod 0.92 mg / Ozanimod 0.92 mg: Participants who received ozanimod in either RPC01-3201 or RPC01-3202 studies receive ozanimod. Participants were administered 0.23 milligram (mg) of Ozanimod capsule (daily) from Day 1 to Day 4 followed by 0.46 mg of Ozanimod (2 capsules of 0.23 mg daily) from Day 5 to Day 7 followed by 0.92 mg of Ozanimod capsule (daily) till discontinuation.
- Ozanimod 0.92 mg / Placebo: Participants who received ozanimod in either RPC01-3201 or RPC01-3202 studies receive placebo orally once daily till discontinuation.
- Placebo / Placebo: Participants who received placebo in either RPC01-3201 or RPC01-3202 studies receive placebo orally once daily till discontinuation in blinded fashion.
Period: Overall Study
Arm/Group | Ozanimod 0.92 mg / Ozanimod 0.92 mg | Ozanimod 0.92 mg / Placebo | Placebo / Placebo
Started (Intent to treat population) | 188 | 188 | 174 (1 participant who was randomized to Placebo/Placebo was actually dosed to Ozanimod 0.92 mg /placebo.)
Safety Population | 188 | 188 | 174
Completed | 96 | 93 | 70
Not Completed | 92 | 95 | 104
Not completed — Withdrawal by Subject | 15 | 13 | 11
Not completed — Study terminated by sponsor | 47 | 44 | 40
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Other reasons | 5 | 12 | 14
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Lack of Efficacy | 11 | 18 | 30
Not completed — Death | 1 | 0 | 0
Not completed — Adverse Event | 13 | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ozanimod 0.92 mg / Ozanimod 0.92 mg | Ozanimod 0.92 mg / Placebo | Placebo / Placebo | Total
Number analyzed (Participants) | 188 | 188 | 174 | 550
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.46 (13.623) | 38.71 (13.916) | 38.68 (13.744) | 39.30 (13.762)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 91 | 83 | 265
  Male | 97 | 97 | 91 | 285
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 14 | 28
  Not Hispanic or Latino | 180 | 175 | 157 | 512
  Unknown or Not Reported | 1 | 6 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  WHITE | 170 | 166 | 153 | 489
  BLACK OR AFRICAN AMERICAN | 3 | 1 | 1 | 5
  AMERICAN INDIAN OR ALASKA NATIVE | 1 | 0 | 1 | 2
  ASIAN | 10 | 13 | 16 | 39
  OTHER | 4 | 4 | 2 | 10
  Unknown or Not Reported | 0 | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve Crohn's Disease Activity Index (CDAI) Score < 150 at Week 52 as Observed
Description: The CDAI is a composite score that is used to measure the clinical activity of Crohn's disease (CD). The CDAI uses a questionnaire with 8 disease activity variables: number of soft/liquid stools, severity of abdominal pain, general well-being, presence of complications, need for antidiarrheal drugs, presence of an abdominal mass, hematocrit, and deviation in body weight. The sub scores of number of soft/liquid stool, severity of abdominal pain (0 [none] to 3 [Severe]), general well-being (0 [well] to 4 [terrible] were summed over the 7 days prior to each visit. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome.
Time Frame: Week 52
Population: Intent-To-Treat population included all randomized participants receiving at least 1dose of investigational product. Only participants with observed cases were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod 0.92 mg / Ozanimod 0.92 mg | Ozanimod 0.92 mg / Placebo | Placebo / Placebo
Number analyzed (Participants) | 147 | 151 | 141
percentage of participants | 44.2 | 33.1 | 35.5
Statistical Analysis 1: Comparison: Ozanimod 0.92 mg / Ozanimod 0.92 mg vs Ozanimod 0.92 mg / Placebo; Test type: Superiority; p = 0.0539, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.59, 95% CI 2-sided [0.99 to 2.55]

2. Primary Outcome: Percentage of Participants With a Simple Endoscopic Score for Crohn's Disease (SES-CD) Score Decrease From Baseline ≥ 50% Based on Observed Cases and Robarts Observed Scores
Description: The SES-CD assessed the degree of inflammation. The SES-CD assesses the following 4 components: size of ulcers, ulcerated surface, affected surface, and presence of narrowing. Each of these components was scored on a scale of 0 (none/unaffected) to 3 (worst). In the SES-CD, each of these 4 components are assessed in the five segments: ileum, right colon, transverse colon, left colon, and rectum. The SES-CD was the sum of the individual scores of each of the components across the five segments. The range of SES-CD scores was 0 - 12 for each segment, and 0 - 60 for the overall SES-CD score, with larger scores indicating greater degree of inflammation. Baseline was defined as the last assessment prior to the start time of the first drug administration if time of measurement is available else the last assessment prior to or on the date of the first drug administration.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod 0.92 mg / Ozanimod 0.92 mg | Ozanimod 0.92 mg / Placebo | Placebo / Placebo
Number analyzed (Participants) | 144 | 154 | 140
percentage of participants | 24.3 | 17.5 | 16.4
Statistical Analysis 1: Comparison: Ozanimod 0.92 mg / Ozanimod 0.92 mg vs Ozanimod 0.92 mg / Placebo; Test type: Superiority; p = 0.1503, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.86 to 2.65]

3. Secondary Outcome: Percentage of Participants With CDAI Reduction From Baseline ≥ 100 Points or CDAI Score <150 at Week 52 as Observed
Description: as for outcome 1
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod 0.92 mg / Ozanimod 0.92 mg | Ozanimod 0.92 mg / Placebo | Placebo / Placebo
Number analyzed (Participants) | 147 | 151 | 141
percentage of participants | 51.0 | 41.7 | 41.1
Statistical Analysis 1: Comparison: Ozanimod 0.92 mg / Ozanimod 0.92 mg vs Ozanimod 0.92 mg / Placebo; Test type: Superiority; p = 0.1121, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.92 to 2.29]

4. Secondary Outcome: Percentage of Participants With Average Daily Abdominal Pain Score ≤1point and Average Daily Stool Frequency ≤ 3 Points With Abdominal Pain and Stool Frequency no Worse Than Baseline at Week 52
Description: Abdominal pain (AP) and stool frequency (SF) clinical remission was defined as average daily abdominal pain score ≤ 1 point, and average daily stool frequency ≤3 times with AP and SF no worse than baseline at Week 12. Participants entered responses in diaries daily. The 7 days entries prior to visit were considered for calculating average AP score and SF. The AP was graded on severity of 0 (none) to 3 (severe) scale and SF was defined number of liquid or soft stools per day.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod 0.92 mg / Ozanimod 0.92 mg | Ozanimod 0.92 mg / Placebo | Placebo / Placebo
Number analyzed (Participants) | 147 | 151 | 141
percentage of participants | 41.5 | 32.5 | 31.9
Statistical Analysis 1: Comparison: Ozanimod 0.92 mg / Ozanimod 0.92 mg vs Ozanimod 0.92 mg / Placebo; Test type: Superiority; p = 0.1163, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.91 to 2.35]

5. Secondary Outcome: Percentage of Participants With With CDAI Score < 150 at Week 52, While Remaining Corticosteroid Free in the 12 Weeks Prior to Week 52 Among All Participants at Maintenance Day 1
Description: as for outcome 4
Time Frame: Week 52
Population: Intent-To-Treat population included all randomized participants receiving at least 1dose of investigational product. Only participants with observed cases remaining corticosteroid free in the 12 weeks prior to Week 52 were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod 0.92 mg / Ozanimod 0.92 mg | Ozanimod 0.92 mg / Placebo | Placebo / Placebo
Number analyzed (Participants) | 93 | 93 | 85
percentage of participants | 48.4 | 34.4 | 45.9
Statistical Analysis 1: Comparison: Ozanimod 0.92 mg / Ozanimod 0.92 mg vs Ozanimod 0.92 mg / Placebo; Test type: Superiority; p = 0.0561, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.78, 95% CI 2-sided [0.98 to 3.20]

6. Secondary Outcome: Percentage of Participants With CDAI Score < 150 at Week 52 in Participants With CDAI Score <150 at Maintenance Day 1
Description: as for outcome 1
Time Frame: Week 52
Population: Intent-To-Treat population included all randomized participants receiving at least 1dose of investigational product. Only participants with observed cases with CDAI score <150 at Maintenance Day 1 were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod 0.92 mg / Ozanimod 0.92 mg | Ozanimod 0.92 mg / Placebo | Placebo / Placebo
Number analyzed (Participants) | 54 | 58 | 56
percentage of participants | 37.0 | 31.0 | 19.6
Statistical Analysis 1: Comparison: Ozanimod 0.92 mg / Ozanimod 0.92 mg vs Ozanimod 0.92 mg / Placebo; Test type: Superiority; p = 0.5061, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.60 to 2.86]

7. Secondary Outcome: Percentage of Participants With Simple Endoscopic Score for Crohn's Disease (SES-CD) ≤ 4 Points and SES-CD Decrease From Baseline ≥ 2points With no SES-CD Subscore > 1 Point at Week 52 Based on Observed Cases
Description: The SES-CD score is a way to measure how severe a person's bowel disease is. It looks at five different parts of the bowel and checks for ulcer size, ulcerated surface, inflamed surface, and stenosis. Each is given a score from 0 to 3 based on how bad the disease is. These scores are then added together for a total score ranging from 0 to 60. Higher scores indicate more severe disease.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod 0.92 mg / Ozanimod 0.92 mg | Ozanimod 0.92 mg / Placebo | Placebo / Placebo
Number analyzed (Participants) | 144 | 154 | 140
percentage of participants | 9.0 | 4.5 | 8.6
Statistical Analysis 1: Comparison: Ozanimod 0.92 mg / Ozanimod 0.92 mg vs Ozanimod 0.92 mg / Placebo; Test type: Superiority; p = 0.1179, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.11, 95% CI 2-sided [0.82 to 5.44]

8. Secondary Outcome: Percentage of Participants With CDAI Score < 150 and SES-CD Decrease From Baseline ≥50% at Week 52 Based on Observed Cases and Robarts Observed Scores
Description: CDAI is a composite score used to measure the clinical activity of Crohn's disease (CD). It assess 8 disease activity variables: number of soft/liquid stools, severity of abdominal pain, general well-being, presence of complications, need for antidiarrheal drugs, presence of an abdominal mass, hematocrit, and deviation in body weight. Sub scores of number of soft/liquid stool, severity of abdominal pain (0 [none] to 3 [Severe]), general well-being (0 [well] to 4 [terrible] were summed over the 7 days prior to each visit. Remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome. SES-CD score is a way to measure how severe a person's bowel disease is. It looks at five different parts of the bowel. Each is given a score from 0 to 3 based on how bad the disease is. These scores are then added together for a total score ranging from 0 to 60. Higher scores indicate more severe disease.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod 0.92 mg / Ozanimod 0.92 mg | Ozanimod 0.92 mg / Placebo | Placebo / Placebo
Number analyzed (Participants) | 144 | 151 | 140
percentage of participants | 19.4 | 11.9 | 12.9
Statistical Analysis 1: Comparison: Ozanimod 0.92 mg / Ozanimod 0.92 mg vs Ozanimod 0.92 mg / Placebo; Test type: Superiority; p = 0.0769, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.78, 95% CI 2-sided [0.94 to 3.39]

9. Secondary Outcome: Percentage of Participants With Average Daily AP Score ≤ 1 Point, and Average Daily Stool Frequency Score ≤ 3 Points With AP and SF no Worse Than Baseline and SES-CD ≤ 4 Points and SES-CD Decrease ≥2 Points With no SES-CD Subscore >1 Point at Week 52
Description: Abdominal pain (AP) and stool frequency (SF) clinical remission was defined as average daily abdominal pain score ≤ 1 point, and average daily stool frequency ≤ 3 times with AP and SF no worse than baseline at Week 12. Participants entered responses in diaries daily. The 7 days entries prior to visit were considered for calculating average AP score and SF. The AP was graded on severity of 0 (none) to 3 (severe) scale and SF was defined number of liquid or soft stools per day. The SES-CD has 4 components size of ulcers, ulcerated surface, affected surface, presence of narrowing. Each component was scored on scale of 0 (none) to 3 (worst). In SES-CD, each of 4 components are assessed in the five segments: ileum, right, transverse, left colon, and rectum. The SES-CD was the sum of the individual scores of each of the components across the five segments. The range of SES-CD scores was 0 - 12 for each segment, and 0 - 60 for overall, with larger scores show greater degree of inflammation.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod 0.92 mg / Ozanimod 0.92 mg | Ozanimod 0.92 mg / Placebo | Placebo / Placebo
Number analyzed (Participants) | 144 | 151 | 140
percentage of participants | 8.3 | 3.3 | 7.9
Statistical Analysis 1: Comparison: Ozanimod 0.92 mg / Ozanimod 0.92 mg vs Ozanimod 0.92 mg / Placebo; Test type: Superiority; p = 0.0623, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.71, 95% CI 2-sided [0.92 to 7.98]

10. Secondary Outcome: Percentage of Participants With CDAI Reduction From Baseline ≥ 100 Points or CDAI Score <150 and SES-CD Decrease From Baseline ≥ 50% at Week 52
Description: as for outcome 8
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod 0.92 mg / Ozanimod 0.92 mg | Ozanimod 0.92 mg / Placebo | Placebo / Placebo
Number analyzed (Participants) | 144 | 151 | 140
percentage of participants | 20.8 | 13.9 | 16.4
Statistical Analysis 1: Comparison: Ozanimod 0.92 mg / Ozanimod 0.92 mg vs Ozanimod 0.92 mg / Placebo; Test type: Superiority; p = 0.1162, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.63, 95% CI 2-sided [0.89 to 3.00]

11. Secondary Outcome: Percentage of Participants With CDAI Reduction From Baseline ≥ 70 Points at Week 52 Based on Observed Cases
Description: CDAI is a composite score used to measure the clinical activity of Crohn's disease (CD). It assess 8 disease activity variables: number of soft/liquid stools, severity of abdominal pain, general well-being, presence of complications, need for antidiarrheal drugs, presence of an abdominal mass, hematocrit, and deviation in body weight. Sub scores of number of soft/liquid stool, severity of abdominal pain (0 [none] to 3 [Severe]), general well-being (0 [well] to 4 [terrible] were summed over the 7 days prior to each visit. Remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod 0.92 mg / Ozanimod 0.92 mg | Ozanimod 0.92 mg / Placebo | Placebo / Placebo
Number analyzed (Participants) | 147 | 151 | 141
percentage of participants | 50.3 | 43.0 | 43.3
Statistical Analysis 1: Comparison: Ozanimod 0.92 mg / Ozanimod 0.92 mg vs Ozanimod 0.92 mg / Placebo; Test type: Superiority; p = 0.2143, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.85 to 2.11]

12. Secondary Outcome: Percentage of Participants With With CDAI Score < 150 at Week 52, While Remaining Corticosteroid Free in the 12 Weeks Prior to Week 52 Among Subjects Using Corticosteroids at Maintenance Day 1
Description: as for outcome 11
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod 0.92 mg / Ozanimod 0.92 mg | Ozanimod 0.92 mg / Placebo | Placebo / Placebo
Number analyzed (Participants) | 146 | 150 | 141
percentage of participants | 39.7 | 29.3 | 30.5
Statistical Analysis 1: Comparison: Ozanimod 0.92 mg / Ozanimod 0.92 mg vs Ozanimod 0.92 mg / Placebo; Test type: Superiority; p = 0.0663, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.58, 95% CI 2-sided [0.97 to 2.57]

13. Secondary Outcome: Percentage of Participants With Mucosal Healing (SES-CD ≤ 4 Points and SES-CD Decrease ≥2 Points With no SES-CD Subscore > 1 Point) and Histologic Improvement Based on Robarts Histologic Index (RHI) at Week 52
Description: as for outcome 2
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod 0.92 mg / Ozanimod 0.92 mg | Ozanimod 0.92 mg / Placebo | Placebo / Placebo
Number analyzed (Participants) | 143 | 151 | 139
percentage of participants | 4.9 | 1.3 | 2.2
Statistical Analysis 1: Comparison: Ozanimod 0.92 mg / Ozanimod 0.92 mg vs Ozanimod 0.92 mg / Placebo; Test type: Superiority; p = 0.0774, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.81, 95% CI 2-sided [0.78 to 18.64]

14. Secondary Outcome: Time to Relapse (an Increase in CDAI Score From Maintenance Day 1 ≥100 Points and CDAI Score >220, SES-CD ≥ 6 [or ≥4 if Isolated Ileal Disease]), and Exclusion of Other Causes of an Increase in Disease Activity Unrelated to Underlying CD
Description: as for outcome 8
Time Frame: Week 52
Population: Intent-To-Treat population included all randomized participants receiving at least 1dose of investigational product.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ozanimod 0.92 mg / Ozanimod 0.92 mg | Ozanimod 0.92 mg / Placebo | Placebo / Placebo
Number analyzed (Participants) | 188 | 188 | 174
days | NA [NA to NA] — Not estimable due to insufficient number of events. | NA [NA to NA] — Not estimable due to insufficient number of events. | NA [NA to NA] — Not estimable due to insufficient number of events.

15. Secondary Outcome: Percentage of Participants With a Crohn's Disease Endoscopic Index of Severity (CDEIS) Decrease From Baseline ≥ 50% at Week 52
Description: CDEIS is an index for determining the severity of Crohn's disease with endoscopic localization to ileum and colon. The CDEIS divides the intestine into 5 segments: rectum, sigmoid and left colon, transverse colon, right colon, and ileum. Four variables are assessed in each segment: the presence of deep ulceration, the presence of superficial ulceration, the percentage of ulcerated surface, and the percentage of surface affected by CD, indicated on 10-cm visual analogue scales. In addition, the presence of ulcerated stenosis and the presence of nonulcerated stenosis are also assessed over the entire intestine. These factors are weighted and summed to calculate the total score ranging from 0- 44, with higher scores indicating more severe disease.
Time Frame: Week 52
Population: Intent-To-Treat population included all randomized participants receiving at least 1dose of investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod 0.92 mg / Ozanimod 0.92 mg | Ozanimod 0.92 mg / Placebo | Placebo / Placebo
Number analyzed (Participants) | 144 | 154 | 140
percentage of participants | 25.7 | 15.6 | 19.3
Statistical Analysis 1: Comparison: Ozanimod 0.92 mg / Ozanimod 0.92 mg vs Ozanimod 0.92 mg / Placebo; Test type: Superiority; p = 0.0308, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.88, 95% CI 2-sided [1.06 to 3.33]

16. Secondary Outcome: Percentage of Participants With CDAI Score < 150 at Week 52 and at ≥ 80% of Visits Between Week 8 and Week 52, Inclusive, in Participants With CDAI Score < 150 at Maintenance Day 1
Description: as for outcome 1
Time Frame: Week 52
Population: Intent-To-Treat population included all randomized participants receiving at least 1dose of investigational product. Participants with with Clinical Remission at Maintenance Day 1 were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod 0.92 mg / Ozanimod 0.92 mg | Ozanimod 0.92 mg / Placebo | Placebo / Placebo
Number analyzed (Participants) | 93 | 93 | 85
percentage of participants | 32.3 | 31.2 | 40.0
Statistical Analysis 1: Comparison: Ozanimod 0.92 mg / Ozanimod 0.92 mg vs Ozanimod 0.92 mg / Placebo; Test type: Superiority; p = 0.8745, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.57 to 1.95]

17. Secondary Outcome: Percentage of Participants With Average Daily Abdominal Pain Score ≤ 1 Point and Average Daily Stool Frequency Score ≤3 Points With Abdominal Pain and Stool Frequency no Worse Than Baseline and SES-CD Decrease From Baseline ≥ 50% at Week 52
Description: Abdominal pain (AP) and stool frequency (SF) clinical remission was defined as average daily abdominal pain score ≤ 1 point, and average daily stool frequency ≤3 times with AP and SF no worse than baseline. Participants entered responses in diaries daily. The 7 days entries prior to visit were considered for calculating average AP score and SF. The AP was graded on severity of 0 (none) to 3 (severe) scale and SF was defined number of liquid or soft stools per day. SES-CD score is a way to measure how severe a person's bowel disease is. It looks at five different parts of the bowel. Each is given a score from 0 to 3 based on how bad the disease is. These scores are then added together for a total score ranging from 0 to 60. Higher scores indicate more severe disease.
Time Frame: Week 52
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod 0.92 mg / Ozanimod 0.92 mg | Ozanimod 0.92 mg / Placebo | Placebo / Placebo
Number analyzed (Participants) | 144 | 151 | 140
percentage of participants | 20.1 | 11.3 | 12.9
Statistical Analysis 1: Comparison: Ozanimod 0.92 mg / Ozanimod 0.92 mg vs Ozanimod 0.92 mg / Placebo; Test type: Superiority; p = 0.0361, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.98, 95% CI 2-sided [1.04 to 3.78]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of Maintenance Study and 90 days after the last dose (up to 731 days). All-cause mortality was collected until 327 weeks.
Description: All-cause mortality, SAEs and Non-SAES were collected for safety population. 1 participant randomized to Placebo/Placebo was actually dosed to Ozanimod 0.92 mg /placebo.
Arm/Group | Ozanimod 0.92 mg / Ozanimod 0.92 mg | Ozanimod 0.92 mg / Placebo | Placebo / Placebo
All-Cause Mortality (participants affected / at risk) | 1/188 | 0/189 | 0/173
Serious Adverse Events (participants affected / at risk) | 12/188 | 17/189 | 19/173
Other Adverse Events (participants affected / at risk) | 27/188 | 43/189 | 34/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ozanimod 0.92 mg / Ozanimod 0.92 mg (N=188) | Ozanimod 0.92 mg / Placebo (N=189) | Placebo / Placebo (N=173)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Microvascular coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 5 | 3 | 8
Enterocolonic fistula (Gastrointestinal disorders) | 1 | 0 | 0
Ileal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 2
Subileus (Gastrointestinal disorders) | 1 | 0 | 0
Liver injury (Hepatobiliary disorders) | 1 | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 2
Appendicitis (Infections and infestations) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 2 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Colonic abscess (Infections and infestations) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ozanimod 0.92 mg / Ozanimod 0.92 mg (N=188) | Ozanimod 0.92 mg / Placebo (N=189) | Placebo / Placebo (N=173)
Crohn's disease (Gastrointestinal disorders) | 14 | 23 | 25
COVID-19 (Infections and infestations) | 11 | 14 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 12 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT03464097/Prot_SAP_000.pdf